CLINICAL TRIAL: NCT05354700
Title: An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) + HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) + Chemotherapy in Patients With Extensive Small Cell Lung Cancer (ES-SCLC)
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of HLX07 Combination Therapy in Patients With Extensive Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-SCLC201
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — HLX07; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX07+HLX10+Chemotherapy (Experimental): HLX07+HLX 10+Chemotherapy (Carboplatin-Etoposide)
  Interventions: Drug: HLX07; Drug: HLX10; Drug: carboplatin and etoposide

INTERVENTIONS:
Drug: HLX07 — HLX07 is a recombinant humanized anti-EGFR monoclonal antibody injection, developed by Shanghai Henlius Biotech, Inc.
Drug: HLX10 — HLX10 is a recombinant humanized anti-PD-1 monoclonal antibody injection, developed by Shanghai Henlius Biotech, Inc.
Drug: carboplatin and etoposide — chemotherapeutics

SUMMARY:
This study is conducted in patients with advanced metastatic small cell lung cancer (SCLC). This study includes a single arm: the patients will receive HLX07 combination therapy with HLX10 and chemotherapy (carboplatin+etoposide) as first-line treatment. All of eligible patients will receive study drug treatment until loss of clinical benefit, unacceptable toxicity, death, withdrawal of informed consent (whichever occurs first, HLX10 treatment up to 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed with ES-SCLC (according to the Veterans Administration Lung Study Group staging system)
* No prior systemic therapy for ES-SCLC
* Major organs are functioning well
* Participant must keep contraception

Exclusion Criteria:

* Histologically or cytologically confirmed mixed SCLC
* Known history of severe allergy to any monoclonal antibody
* Known hypersensitivity to carboplatin or etoposide
* Pregnant or breastfeeding females
* Patients with a known history of psychotropic drug abuse or drug addiction
* Patients who have other factors that could lead to the early termination of this study based on the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-29 (Estimated); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-05-29 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate by investigator assessment per RECIST 1.1
PFS | Up to 2 years
  Progression-free survival by investigator assessment per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided